CLINICAL TRIAL: NCT06697301
Title: A Multicenter, Randomized, Double-Blind, Active Comparator-Controlled, Adaptive Phase 2/3 Study to Evaluate the Safety and Efficacy of EIK1001 and Pembrolizumab Versus Placebo and Pembrolizumab as First-Line Therapy in Participants With Advanced Melanoma (TeLuRide-006)
Brief Title: Safety and Efficacy of EIK1001 in Combo With Pembro Versus Placebo and Pembro as First-Line Therapy in Patients With Advanced Melanoma.
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eikon Therapeutics (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EIK1001-006; KEYNOTE-G04 (Other: Merck Sharp & Dohme LLC); MK-3475-G04 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Advanced Melanoma
Keywords: Metastatic; Advanced
MeSH Terms: conditions — Neoplasm Metastasis | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Active Comparator): Participants in this arm will receive Placebo and Standard of Care (Pembrolizumab).
  Interventions: Drug: Pembrolizumab (KEYTRUDA® )
- Arm 2 (Experimental): Participants in this arm will receive EIK1001 (selected dose 1) + Standard of Care (Pembrolizumab).
  Interventions: Drug: EIK1001; Drug: Pembrolizumab (KEYTRUDA® )
- Arm 3 (Experimental): Participants in this arm will receive EIK1001 (selected dose 2) + Standard of Care (Pembrolizumab).
  Interventions: Drug: EIK1001; Drug: Pembrolizumab (KEYTRUDA® )

INTERVENTIONS:
Drug: EIK1001 — EIK1001 is a Toll-like receptor 7/8 (TLR 7/8) dual agonist.
  Arms: Arm 2; Arm 3
Drug: Pembrolizumab (KEYTRUDA® ) — Pembrolizumab is a PD-1 inhibitor.

SUMMARY:
The study is for patients with advanced melanoma who are eligible for standard therapy with Pembrolizumab.

DETAILED DESCRIPTION:
This is a Multicenter, Randomized, Double-Blind, Active Comparator-Controlled, Adaptive Phase 2/3 Study to Evaluate the Safety and Efficacy of EIK1001 and Pembrolizumab Versus Placebo and Pembrolizumab as First-Line Therapy in Participants with Advanced Melanoma. The study includes dose optimization and expansion parts.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion in this study, participants must:

* Be ≥ 18 years of age on the day of signing of informed consent.
* Have a life expectancy of at least 3 months.
* Have histologically or cytologically confirmed Stage 3 (unresectable) or Stage 4 metastatic melanoma per AJCC 8th ed. and be eligible for standard therapy with pembrolizumab.
* Have at least 1 lesion with measurable disease at Baseline by CT or MRI according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 by assessment of local site Investigator/radiologist.
* Have known BRAF V600 mutation status or consent to BRAF V600 mutation testing per local institutional standards during the screening period
* Have completed prior radiotherapy at least 2 weeks prior to study treatment administration.
* Have an ECOG Performance Status of 0 to 1.
* Have adequate organ and marrow function as defined by normal CBC, coagulation, serum chemistry and liver function tests on specimens collected within 10 days of treatment start.
* Have a negative serum pregnancy test within 72 hours prior to receiving the first dose of study medication (applies to women of childbearing potential [WOCBP]).
* Be willing to use either 2 adequate methods of contraception, 1 adequate method plus a hormonal method of contraception, or be willing to abstain from heterosexual activity throughout the study (Visit 1 to 120 days after the last dose of study therapy; applies to WOCBP who are not menopausal for > 2 years, post-hysterectomy/oophorectomy, or surgically sterilized).
* Agree to use an approved adequate contraceptive method throughout the study (Visit 1 to 120 days after the last dose of study therapy; applies to sexually active male participants with a partner who is WOCBP).
* Be willing and able to provide written, informed consent for the study.

Exclusion Criteria:

A participant is excluded from the study if any of the following criteria apply:

* Has melanoma of ocular origin.
* Is currently enrolled in or has recently participated in a study of an IMP and received an IMP within 4 weeks or 5 half-lives (whichever is shorter) of administration of EIK1001 or placebo.
* Prior to the 1St dose of EIK1001 or placebo, the prospective participant has received systemic therapy for advanced melanoma.
* Note: prior adjuvant or neoadjuvant melanoma therapies (such as anti-PD-1 or anti CTLA 4 therapies or BRAF/MEK inhibitors) are permitted if all related AEs have either returned to Baseline or stabilized, with a minimum of 6 months between the last dose of prior therapy and documented disease progression.
* Experienced a ≥ Grade 3 AE while receiving prior anti PD 1 therapy.
* Has had major surgery (< 3 weeks prior to the first dose).
* Has received a live-virus vaccination within 30 days of the first dose of study treatment.
* Has a known history of prior malignancy, unless the participant has undergone potentially curative therapy with no evidence of disease recurrence for 5 years.
* Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate if they are clinically stable for at least 4 weeks with no evidence of new or enlarging brain metastases. There must be no need for immunosuppressive doses of glucocorticoids for at least 2 weeks prior to study treatment administration.
* There is a mean resting QTcF > 470 ms on triplicate electrocardiograms.
* There is active autoimmune disease that has required systemic treatment in the past 2 years. The following autoimmune conditions are permitted: Type 1 diabetes, hypothyroidism (on hormone replacement), or- vitiligo, psoriasis and alopecia as long as no systemic treatment is required.
* There is either chronic treatment with systemic steroids, other immunosuppressive medication, or either of these has been administered within 14 days of start of study treatment.
* Note: Participants with asthma that require intermittent use of bronchodilators, inhaled steroids, or local steroid injections are eligible. Steroid replacement for adrenal insufficiency is also permitted.
* There is a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/ interstitial lung disease.
* There are any active infections requiring therapy.
* There is uncontrolled human immunodeficiency virus (HIV) infection. HIV-infected participants with well-controlled HIV may enroll.
* There is a positive test result for hepatitis B virus (HBV) or HCV indicating presence of virus (it is expected that all participants will have been serologically tested for hepatitis B in advance of this study, with HBsAG, anti-HBc IgG, and anti-HBs as per ASCO 2020 Provisional Clinical Opinion [PCO] on universal Serologic testing for hepatitis B at the onset of anticancer therapy; screening should also include an anti-HCV test prior to start of cancer treatment:
* There is a history or clinical evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study or interfere with the participant's participation for the full duration of the study
* Known psychiatric or substance abuse disorder that would interfere with cooperation with study requirements.
* There is a known history of regular illicit drug use and/or recent history (within the last year) of substance abuse (including alcohol).
* Participant is pregnant, breastfeeding, or planning to conceive or father children within the projected duration of the study.
* Participant is currently receiving medications known to be strong inhibitors or inducers of CYP3A4 and CYP1A2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 740 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | up to 5 years
  Progression-free survival (PFS) is defined as the time from the date of randomization to documented progressive disease per RECIST 1.1 by BICR or death due to any cause, whichever occurs first.
Overall survival (OS) | up to 5 years
  Overall survival (OS) defined as the time from randomization to death due to any cause.
Objective Response (OR) (Dose Optimization Only) | up to 5 years
  Objective Response (OR; defined as participants who demonstrate confirmed complete response [CR] or partial response [PR] by Response Evaluation Criteria in Solid Tumors [RECIST] version 1.1 as assessed by the Investigator) (Dose Optimization Only).
Adverse Events (AEs) (Dose Optimization Only) | up to 2.5 years
  Adverse events (AEs), and discontinuation of study treatment due to an AE (Dose Optimization Only). An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment.

SECONDARY OUTCOMES:
Adverse Events (AEs) and Discontinuation of study treatment due to any AE. | up to 2.5 years
  Adverse events (AEs), and discontinuation of study treatment due to any AE. An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Objective Response (OR) | up to 5 years
  Objective response (OR) is defined as the participants who demonstrate confirmed response (CR) or partial response (PR) according to RECIST 1.1 by BICR.
Duration of Response (DOR). | up to 5 years
  Duration of Response (DOR) is defined as the time from the first documented evidence of complete response (CR) or partial response (PR) until disease progression or death due to any cause, whichever occurs first according to RECIST 1.1 by BICR.
Progression Free Survival (PFS) | up to 5 years
  Progression Free Survival (PFS) according to RECIST 1.1 by Investigator.
Objective Response (OR) | up to 5 years
  Objective Response (OR) according to RECIST 1.1 by Investigator.
Duration of Response (DOR) | up to 5 years
  Duration of Response (DOR) according to RECIST 1.1 by Investigator
Duration of Response (DOR) (Dose Optimization Only). | up to 5 years
  Duration of Response (DOR) per RECIST 1.1 by Investigator (Dose Optimization Only).
Progression-free survival (PFS) per RECIST 1.1 by Investigator (Dose Optimization Only). | up to 5 years
  Progression-free survival (PFS) per RECIST 1.1 by Investigator (Dose Optimization Only).
Overall survival (OS) (Dose Optimization Only) | up to 5 years
  Overall survival (OS) defined as the time from randomization to death due to any cause (Dose Optimization Only).

CONTACTS AND LOCATIONS:
Overall Officials: Etah Kurland, Study Director — Eikon Therapeutics; Muaz Sadeia, Study Director — Eikon Therapeutics
Locations (77):
- United States (11):
  - Ironwood Cancer & Research Centers, Chandler, Arizona
  - Genesis Cancer and Blood Institute, Hot Springs, Arkansas
  - Helios Clinical Research, Los Angeles, California
  - Providence Medical Foundation, Santa Rosa, California
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Bioresearch Partner, Hialeah, Florida
  - The Center for Cancer and Blood Disorders, Bethesda, Maryland
  - MidAmerica Cancer Care, Kansas City, Missouri
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Gabrail Cancer Center Research LLC, Canton, Ohio
  - University of Pittsburgh Medical Center(UPMC)-Hillman Cancer Center, Pittsburgh, Pennsylvania
- Australia (4):
  - Cancer Care Wollongong, Wollongong, New South Wales
  - Icon Cancer Centre Chermside, Chermside, Queensland
  - Southern Adelaide Local Health Network Incorporated Flinders Medical Centre, Bedford Park, South Australia
  - Eastern Health, Box Hill, Victoria
- Universitätsklinikum Graz, Graz, Styria, Austria
- Belgium (5):
  - Universitair Ziekenhuis Antwerpen, Edegem, Antwerpen
  - Cliniques Universitaires Saint-Luc, Brussels, Brussels Capital
  - Centre Hospitalier Universitaire Universite Catholique de Louvain - Site Godinne, Yvoir, Namur
  - Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven, Vlaams Brabant
  - Algemeen Ziekenhuis Groeninge - Campus Kennedylaan, Kortrijk, West-Vlaanderen
- Sunnybrook Research Ins<tute, Toronto, Ontario, Canada
- Czechia (2):
  - Masaryk Memorial Cancer Institute, Brno, Brno
  - University Hospital Hradec Kralove, Sokolov, Hradce Kralove
- Denmark (2):
  - Aarhus Universitetshospital, Aarhus, Central Jutland
  - Aalborg University Hospital, Aalborg, Nord Jutland
- Finland (3):
  - Oulu University Hospital, Oulu, Oulu
  - Tampere University Hospital, Tampere, Pirkanmaa
  - Helsinki University Hospital, Helsinki, Uusimaa
- France (4):
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite, Auvergne-Rhône-Alpes
  - Centre Hospitalier Universitaire Grenoble Alpes, La Tronche, Isère
  - Hôpital La Timone, Marseille, Marseille
  - CHU Rouen, Rouen, Rouen
- Germany (8):
  - Universitätsmedizin Mannheim, Mannheim, Baden-Wurttemberg
  - Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg
  - Universitat Leipzig, Saxony, Leipzig
  - Elbe Kliniken Stade-Buxtehude, Buxtehude, Lower Saxony
  - Johannes Wesling Klinikum Minden, Minden, North Rhine-Westphalia
  - University of Mainz Medical Center, Mainz, RLP
  - Universitätsklinikum Schleswig-Holstein - Campus Kiel, Kiel, Schleswig-Holstein
  - Universitätsklinikum Schleswig-Holstein - Campus Lübeck, Lübeck, Schleswig-Holstein
- Israel (4):
  - Soroka medical center, Beersheba, Be'er Sheva
  - Rabin Medical Center, Petah Tikva, Petach Tikva
  - Ella Lemelbaum Institute for Immuno-Oncology and Melanoma, Ramat Gan, Ramat Gan
  - Tel Aviv Medical Center, Tel Aviv, Tel Aviv
- Humanitas Gavazzeni Bergamo, Bergamo, Province of Bergamo, Italy
- New Zealand (2):
  - Christchurch Public Hospital, Christchurch, Christchurch
  - Auckland City Hospital, Auckland, New Zealand
- Norway (2):
  - Nordland Hospital Trust, Bodø, Bodø
  - Oslo University Hospital - The Norwegian Radium Hospital, Oslo, Oslo County
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne, Gdansk, Gdańsk
  - Prezychodnia Lekarska KOMED Roman Karaszewski, Konin, Konin
  - Mazowiecki Szpital Wojewódzki, Siedlckie Centrum Onkologii, Siedlce, Siedlce
- Hospital da Luz Lisboa, Lisbon, Lisbon District, Portugal
- Military Medical Academy- Department of Oncology, Belgrade, Belgrade, Serbia
- South Africa (5):
  - Cancercare Port Elizabeth - Langenhoven Drive Oncology Centre, Port Elizabeth, Eastern Cape
  - University of Pretoria, Steve Biko Academic Hospital, Pretoria, Gauteng
  - The Medical Oncology Centre of Rosebank, Saxonwold, Gauteng
  - Cape Town Oncology Trials, Cape Town, Western Cape
  - TASK Eden, George Central, Western Cape
- Spain (11):
  - Hospital Universitari Dexeus, Barcelona, Barcelona
  - Vall d' Hebron Institute of Oncology, Barcelona, Barcelona
  - Hospital Universitario Lucus Augusti, Lugo, Galicia
  - Institut Català d'Oncologia Girona (ICO Girona), Girona, Girona
  - University Hospital of Jerez, Jerez de La Frontera (Cádiz), Jerez de La Frontera (Cádiz)
  - GenesisCare Madrid - Hospital San Francisco de Asís, Madrid, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid, Madrid
  - Hospital 12 de Octubre, Usera, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga, Málaga
  - IVO - Fundacion Instituto Valenciano de Oncologia, Valencia, Valencia
  - INCLIVA Instituto de Investigación Sanitaria, Valencia, Valencia
- Sweden (2):
  - Gävle Sjukhus, Gävle, Gävleborg County
  - Karolinska University Hospital, Stockholm, Södermanland County
- Switzerland (2):
  - Universitätsspital Zürich, Zurich, Canton of Zurich
  - Kantonsspital Graubünden, Chur, Chur
- United Kingdom (2):
  - Guy's and St Thomas' NHS Foundation Trust, London, England
  - Sarah Cannon Research Institute London, London, England